CLINICAL TRIAL: NCT02433249
Title: Enhancing Motivation for Physical Activity to Reduce the Risk of Falls Among Community-Dwelling Older Adults: A Wellness Intervention.
Brief Title: Developing a Intervention to Enhance Motivation for Physical Activities Known to Reduce Fall Risk
Acronym: ReadySteady
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1402S47802
Record Dates: First submitted 2015-02-19; First posted 2015-05-04 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Accidental Falls; Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 Physical Activity (Active Comparator): Small groups (4-7 people) meeting in community centers weekly for 90 minutes, over the course of 8 weeks. Curricula for meetings are manualized and include introducing and practicing Otago exercises, progressed according to individual capacity and preference, as well as falls prevention. All participant receive Fitbit Ones and are asked to use them on a daily basis.
  Interventions: Behavioral: 1 Physical Activity
- 2 Interpersonal Motivation (Experimental): Small groups (4-7 people) meeting in community centers weekly for 90 minutes, over the course of 8 weeks. Curricula for meetings are manualized and include introducing and practicing Otago exercises, progressed according to individual capacity and preference, as well as falls prevention. The interventionist also facilitates discussions addressing the interpersonal motivational intervention content. All participant receive Fitbit Ones and are asked to use them on a daily basis: Fitbit Ones are included in weekly discussions.
  Interventions: Behavioral: 1 Physical Activity; Behavioral: Interpersonal Motivation
- 3.Intrapersonal Motivation (Experimental): Small groups (4-7 people) meeting in community centers weekly for 90 minutes, over the course of 8 weeks. Curricula for meetings are manualized and include introducing and practicing Otago exercises, progressed according to individual capacity and preference, as well as falls prevention. The interventionist also facilitates discussions addressing the intrapersonal motivational intervention content. All participant receive Fitbit Ones and are asked to use them on a daily basis: Fitbit Ones are included in weekly discussions.
  Interventions: Behavioral: 1 Physical Activity; Behavioral: Intrapersonal Motivation
- 4.Full Intervention (Experimental): Small groups (4-7 people) meeting in community centers weekly for 90 minutes, over the course of 8 weeks. Curricula for meetings are manualized and include introducing and practicing Otago exercises, progressed according to individual capacity and preference, as well as falls prevention. The interventionist also facilitates discussions addressing the intrapersonal and interpersonal motivational intervention content. All participant receive Fitbit Ones and are asked to use them on a daily basis: Fitbit Ones are included in weekly discussions.
  Interventions: Behavioral: 1 Physical Activity; Behavioral: Interpersonal Motivation; Behavioral: Intrapersonal Motivation

INTERVENTIONS:
Behavioral: 1 Physical Activity — Fall reducing strength (5), balance (12) and flexibility (4) exercises as well as walking. Participants were also given a Fitbit One with instructions on how to use
  Other Names: Otago
Behavioral: Interpersonal Motivation — Strategies used to support Interpersonal motivational targets include: a) discuss and model ways to provide and receive more support for physical activity, b) identify environmental barriers to being physically active, c) problem-solve environmental and social barriers to being physically active, d) use and create new resources that support physical activity behavior
  Arms: 2 Interpersonal Motivation; 4.Full Intervention
Behavioral: Intrapersonal Motivation — Strategies used to support intrapersonal motivation included a) use of the goal attainment scale, b) facilitating the formation of action plans, c) identify and problem solve personal barriers to being active, d) identify satisfying aspects of being active, e) self-evaluate physical activity patterns and progress.
  Arms: 3.Intrapersonal Motivation; 4.Full Intervention

SUMMARY:
The purpose of this pilot study is to develop an intervention, based on empirical evidence and health-related behavioral change theory, to enhance motivation for engaging in fall-reducing physical activities.

DETAILED DESCRIPTION:
The intervention being developed, Ready~Steady, combines 3 components; a) interpersonal motivation, b) intrapersonal motivation, and c) physical activity. Theoretical concepts from the wellness motivation theory are (a) translated into intervention strategies; and (b) operationalized as variables to form a basis for evaluating this intervention. The overall objective is to advance the development of Ready~Steady by assessing the impact of its motivation components.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 years, level of physical activity (strength training and aerobic) below national recommendations

Exclusion Criteria:

* Dementia, recent injury or surgery, unable to participate in light-moderately intense exercise

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in self-reported physical activity behavior | Baseline; 1 week post; 6 months post
  Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire
Change in objectively measured physical activity behavior | Baseline; 1 week post; 6 months post
  Accelerometers built in to Fitbit Ones

SECONDARY OUTCOMES:
Change in functional strength and balance | Baseline; 1 week post; 6 months post
  Short Physical Performance Battery
Change in functional strength and balance | Baseline; 1 week post; 6 months post
  Timed Up and Go
Change in the number of community resources used for physical activity | Baseline; 1 week post; 6 months post
  Number of community resources identified and used: 2 item survey
Change in social support for fall-reducing physical activities | Baseline; 1 week post; 6 months post
  Social support for exercise: Survey
Change in readiness | Baseline; 1 week post; 6 months post
  Index of Readiness
Change in self-regulation | Baseline; 1 week post; 6 months post
  Index of Self-Regulation
Change in self-reported lower extremity function | Baseline; 1 week post; 6 months post
  Neuro-QOL SF v1.0 - LEx Fnct (Mobility)
Change in self-reported ability to participate in social activities | Baseline; 1 week post; 6 months post
  PROMIS SF v2.0 - Ability to Participate Social 4a

OTHER OUTCOMES:
Technology acceptability and utility | 1 week post; 6 months post
  10 item survey addressing wearable technology's learnability, utility and role in supporting individual motivation

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan K McMahon, PhD, Principal Investigator — University of Minnesota

REFERENCES:
- [Background] McMahon S, Vankipuram M, Hekler EB, Fleury J. Design and evaluation of theory-informed technology to augment a wellness motivation intervention. Transl Behav Med. 2014 Mar;4(1):95-107. doi: 10.1007/s13142-013-0221-4. PMID 24653780
- [Background] McMahon S, Fleury J. Wellness in older adults: a concept analysis. Nurs Forum. 2012 Jan-Mar;47(1):39-51. doi: 10.1111/j.1744-6198.2011.00254.x. PMID 22309381
- [Background] Perez A, Fleury J. Wellness motivation theory in practice. Geriatr Nurs. 2009 Mar-Apr;30(2 Suppl):15-20. doi: 10.1016/j.gerinurse.2009.02.006. No abstract available. PMID 19345859
- [Background] McMahon S, Talley KM, Wyman JF. Older people's perspectives on fall risk and fall prevention programs: a literature review. Int J Older People Nurs. 2011 Dec;6(4):289-98. doi: 10.1111/j.1748-3743.2011.00299.x. PMID 22078019
- [Derived] McMahon SK, Lewis B, Oakes JM, Wyman JF, Guan W, Rothman AJ. Examining Potential Psychosocial Mediators in a Physical Activity Intervention for Older Adults. West J Nurs Res. 2020 Aug;42(8):581-592. doi: 10.1177/0193945919871697. Epub 2019 Aug 30. PMID 31470769
- [Derived] McMahon SK, Lewis B, Oakes JM, Wyman JF, Guan W, Rothman AJ. Assessing the Effects of Interpersonal and Intrapersonal Behavior Change Strategies on Physical Activity in Older Adults: a Factorial Experiment. Ann Behav Med. 2017 Jun;51(3):376-390. doi: 10.1007/s12160-016-9863-z. PMID 28188585
- [Derived] McMahon SK, Lewis B, Oakes M, Guan W, Wyman JF, Rothman AJ. Older Adults' Experiences Using a Commercially Available Monitor to Self-Track Their Physical Activity. JMIR Mhealth Uhealth. 2016 Apr 13;4(2):e35. doi: 10.2196/mhealth.5120. PMID 27076486